CLINICAL TRIAL: NCT03741959
Title: Rehabilitation of Postural Abnormalities in Parkinson's Disease: a Single-blind, Randomised Controlled Trial
Brief Title: Rehabilitation of Postural Abnormalities in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Head of UOC Neurorehabilitation, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REMoVE Study
Record Dates: First submitted 2018-09-01; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Parkinson Disease
Keywords: postural defect
MeSH Terms: conditions — Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment. Single-blind RCT with two parallel group
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded. Patients will be specifically asked not to discuss their treatment during assessments. Examiner will be requested to inform the research coordinator if he will discover to which group a patient belonged, and they will periodically be questioned by the coordinator about this.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will undergo three groups of exercises: 1) active self-correction exercises (20 minutes) defined as the best possible trunk alignment the patient can achieved in the three-dimensional planes; 2) passive and active trunk stabilization exercises (20 minutes) to improve trunk biomechanical constraint and to counteract the evolution of the misalignment; 3) functional tasks (20 minutes) defined as functional exercises to train the automatic response to maintain the best alignment through the broadest possible range of challenging activities (Romano2015).Training will consist of individualized treatment 60 mins/day, 2 days/week, for 5 consecutive weeks.
  Interventions: Procedure: Experimental group
- Control (Active Comparator): The control group will undergo strengthening exercises and gait training as the usual practice in Parkinson Disease. Training will consist of individualized treatment 60 mins/day, 2 days/week, for 5 consecutive weeks (Bartolo et. al., 2010).
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Experimental group — Active self-correction exercises (20 minutes) to achieve the best possible trunk alignment the patient can achieve in the three-dimensional planes using visual, proprioceptive and EMG feedbacks.
  Passive and active trunk stabilization exercises (20 minutes) to improve trunk biomechanical constraint Functional tasks (20 minutes) defined as functional exercises to train the automatic response to maintain the best alignment through the broadest possible range of challenging activities (Romano2015).
  Arms: Experimental
Procedure: Control group — Training consisted of passive and active trunk mobilization (10 minutes) followed by muscle stretching, and strengthening exercises, and gait training (50 minutes)(Bartolo et. al., 2010).
  Arms: Control

SUMMARY:
Postural abnormalities (PA) are drug refractory complications in patients with Parkinson's disease (PD) leading to pain, imbalance, gait disorders and fall-related injuries. It ultimately affects the quality of life and the hospitalisation risk. the literature on treatment outcomes is scant. Rehabilitation is the cornerstone in the management of PD patients, especially for drug-refractory complications. However, the current efforts are only partially able to resolve PA in PD. Despite differences in methodologies, the few rehabilitative studies support the benefits of trunk rehabilitation in PD with PA. Priorities for future research include well-design rehabilitation studies on a large population. The early detection and early rehabilitation of PA might avoid fixed irreversible deformities and reduce the complications that can accompany them. It ultimately might improve the quality of life, reduce the risk of fall-related injuries and hospitalisation rate. A single-blind single-blind Randomised Controlled Trial (RCT) will evaluate the effects of trunk rehabilitation on PA severity, function and disability in outpatients with Parkinson Disease and postural abnormalities.

DETAILED DESCRIPTION:
This RCT with two parallel group will be conducted according to the tenets of the Declaration of Helsinki, the guidelines for Good Clinical Practice, and the Consolidated Standards of Reporting Trials (CONSORT).

The target population will be patients with Parkinson Disease who attend to the Neurorehabilitation Unit (AOUI Verona) and the Unità Operativa Complessa (UOC) Neurology ward (AOUI Verona) where they will be assessed for eligibility.

Who satisfied inclusion and exclusion criteria were randomly allocated in one of two groups, the experimental group and control group. Each patient will undergo rehabilitation.

Before the start of the study authors designed the experimental and the control group protocols. Two physiotherapists, one for each group, carried out the rehabilitation procedures. Patients of both groups received 10 individual sessions (60 min/session, 2 sessions/week, five consecutive weeks). Treatments will be performed in the rehabilitative gym of the G.B. Rossi University Hospital Neurological Rehabilitation Unit.

For the statistical analysis, an intention to treat analysis will be used. Descriptive statistics included means, standard deviation and graphs. The Shapiro-Wilk test will be used to test data distribution. Parametric or non-parametric tests will be used for inferential statistics, accordingly. The T-Test for unpaired data (or the Mann-Whitney test) will be used for testing between-group differences at T0 and T1. For this purpose, the changes of the score (Δ) between T0-T1 will be computed. The T-Test for paired data (or Wilcoxon signed rank tests) will be used to compare within-group changes over time. The level of significance was set p<0.05. Software statistics SPSS 20.0 (IBM Statistical Package for Social Science (SPSS) Statistics for Windows, Version 20.0, Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Age higher than 18 years old:
* A medical diagnosis of PD confirmed according to the Movement disorders criteria;
* PS defined as at least 10 degrees of lateral trunk flexion that can be reduced by passive mobilization or supine positioning (PS≥10) (Doherty et. al., 2011);
* Camptocormia defined as a flexion (at least 5°) in the sagittal plane originating in the thoracolumbar spine, (classified as upper and lower), manifesting during standing and walking and completely subside in recumbent position (Pandey et. al., 2016);
* Hoehn & Yahr (H&Y) stage <4 in "ON" medication phase.
* Informed consent to participate in the study

Exclusion Criteria:

* Severe dyskinesia or "on-off" fluctuations;
* PD medication modification in the 3 months preceding enrollment into the study;
* Need for assistive devices to rise from a chair or bed; somatic sensation deficits involving the legs;
* Vestibular disorders or paroxysmal vertigo; other neurological, orthopaedic or cardiovascular co-morbidities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the degrees of trunk deviation in the sagittal and coronal plane. | Pre-treatment, after 5 weeks, at 1 month-follow-up and 4-month follow-up
  Changes in the degree of trunk deviation in the sagittal and coronal plane will be assessed using a wall goniometer in standing position.

SECONDARY OUTCOMES:
Changes in Gait speed (cm/sec) | Pre-treatment, after 5 weeks, at 1 month-follow-up and 4-month follow-up
  Changes in gait speed will be assessed using the Gait Rite System. It is a computerized walkway providing temporal spatial gait analysis.
Changes in the Percentage Difference of Sway (PDS) | Pre-treatment, after 5 weeks, at 1 month-follow-up and 4-month follow-up
  The PDS computed for sway velocity in the eyes open (eo) and eyes closed (ec) conditions. A ratio close to zero or negative indicates that the magnitude of body sway is similar or smaller in the ec than in the eo condition . On the contrary, positive values reflect a larger sway in the ec than in the eo condition.
Changes in the Unified Parkinson's Disease Rating Scale (UPDRS) | Pre-treatment, after 5 weeks, at 1 month-follow-up and 4-month follow-up
  It is a comprehensive assessment designed to monitor the burden and the extent of Parkinson Disease across the longitudinal disease course and provides a clinical end-point in clinical trials. It consists of four sections with a total summed score. Each item have 5 response options (0=normal; 4=severe symptoms/signs). The higher= greater impact of PD symptoms.
  The Unified Parkinson's Disease Rating Scale - part III (UPDRS III) subscale will be used to measure changes in the motor disability (score range, 0-33; the higher=worse symptoms).
Changes in the Parkinson's Disease Questionnaire (PDQ-8) | Pre-treatment, after 5 weeks, at 1 month-follow-up and 4-month follow-up
  The PDQ-8 contains eight of the original 39 items of the PDQ-39; one item selected from each of the 8 scales (mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communications and bodily discomfort). It provides a reliable measure of overall health status and is ideal for studies in which a shorter questionnaire is preferred. Each question is scored from 0-4 points and the scores are summed. the summed scores are then divided by total possible score and given as a percentage score out of 100 (Score range, 32-100; the higher worse health status)
The number of falls | Pre-treatment, after 5 weeks, at 1 month-follow-up and 4-month follow-up
  Number of falls occured in the previous month.
Changes in the Mini Balance Evaluation System test (Mini BESTest) | Pre-treatment, after 5 weeks, at 1 month-follow-up and 4-month follow-up
  It is a clinical balance assessment tool to target and identify 4 different balance control systems (anticipatory postural adjustments, reactive postural control, sensory orientation, dynamic gait) so that specific rehabilitation approaches can be designed. It is a 14-item test scored on a 3-level ordinal scale (0-2). Total score range 0-32; the higher= better performance.
Changes in the Numeric Pain Rating Scale (NPRS) | Pre-treatment, after 5 weeks, at 1 month-follow-up and 4-month follow-up
  A numeric rating scale to measure the amount of pain that a patient feels ranges across a continuum from none (0) to an extreme amount of pain (10). Total score range 0-10; the higher= worse performance.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tinazzi, PhD, Study Chair — Universita di Verona
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartolo M, Serrao M, Tassorelli C, Don R, Ranavolo A, Draicchio F, Pacchetti C, Buscone S, Perrotta A, Furnari A, Bramanti P, Padua L, Pierelli F, Sandrini G. Four-week trunk-specific rehabilitation treatment improves lateral trunk flexion in Parkinson's disease. Mov Disord. 2010 Feb 15;25(3):325-31. doi: 10.1002/mds.23007. PMID 20131386
- [Result] Doherty KM, van de Warrenburg BP, Peralta MC, Silveira-Moriyama L, Azulay JP, Gershanik OS, Bloem BR. Postural deformities in Parkinson's disease. Lancet Neurol. 2011 Jun;10(6):538-49. doi: 10.1016/S1474-4422(11)70067-9. Epub 2011 Apr 22. PMID 21514890
- [Derived] Gandolfi M, Tinazzi M, Magrinelli F, Busselli G, Dimitrova E, Polo N, Manganotti P, Fasano A, Smania N, Geroin C. Four-week trunk-specific exercise program decreases forward trunk flexion in Parkinson's disease: A single-blinded, randomized controlled trial. Parkinsonism Relat Disord. 2019 Jul;64:268-274. doi: 10.1016/j.parkreldis.2019.05.006. Epub 2019 May 3. PMID 31097299